CLINICAL TRIAL: NCT05697172
Title: Neuromodulation of Circuits Underlying Repetitive Negative and Self-Referential Thinking in Depression: An Early Feasibility Study Employing Transcranial Focused Ultrasound
Brief Title: Low Intensity Ultrasound Neuromodulation of Repetitive Negative Thinking In Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2021-011
Record Dates: First submitted 2022-11-11; First posted 2023-01-25 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder
Keywords: Repetitive Negative Thinking; Low-Intensity Focused Ultrasound; Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: An exploratory hypothesis is that stimulation of anteromedial structures of the telencephalic cortex of the right hemisphere and their connections with subcortical structures will lead to detectable attenuation of RNT in high RNT depressed individuals. In this study, the investigators will use a double-blind, randomized cross-over design employing either tfUS or sham stimulation. The proposed design parsimoniously follows the approved pilot study supported by the Center of Biomedical Research Excellence grant NeuroMAP (P20GM121312), in which the investigators will characterize neural circuits associated to RNT.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A sound proof material will be employed to deliver sham stimulation. The operator of the device will be unblinded to the type of intervention (verum vs sham). Participant, assessment team including raters, and staff responsible for evaluation of psychiatric and neurological status will be blind to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Low Intensity Focused Ultrasound (LIFU) (Experimental): An 80-second train of 20-millisecond bursts of ultrasound (0.5 MHz), repeated every 200 milliseconds (400 bursts). Acoustic simulations will be performed with the k-Wave Matlab Toolbox to individually confirm the estimated total energy delivered during sonication and verify tissue temperature increases are <1°C, decreasing actual Power/Channel values if necessary. We estimate a 75% tissue attenuation of energy when the ultrasound wave reaches its target, therefore we will set the free-field Intensity Spatial-Peak Pulse-Average (ISPPA) at 9.04 Watt /cm2 or 518 kPascal (to achieve 2.26 Watt/cm2 derated ISPPA).
  Interventions: Other: Low-intensity focused ultrasound
- Sham LIFU (Sham Comparator): Identical parameters of sonication and positioning procedures as those in the Active LIFU arm will be employed, but a Sorbothane(R) film will be interposed between the transducer and the subject's scalp.
  Interventions: Other: Low-intensity focused ultrasound

INTERVENTIONS:
Other: Low-intensity focused ultrasound — 80-second stimulus with an estimated tissue ISSPA=2.26 W/cm2, with (sham) or without (verum) interposition of Sorbothane film

SUMMARY:
The investigators propose to use low-intensity transcranial focused ultrasound (LIFU), a novel neuromodulation method, to probe the causal involvement of individually defined components of an anteromedial brain circuit in the processing of self-referential thoughts, and the production of repetitive negative thinking (RNT), a prominent transdiagnostic manifestation with adverse clinical consequences. The investigators hypothesize that real vs. sham low-intensity sonication of individually-defined anteromedial structures connecting medial orbitofrontal and anterior cingulate cortices with ventral striatum and anterior thalamus will show reduced initiation or maintenance of RNT as measured by (1) Brief State Rumination Inventory (BSRI) scores and distress associated to repetitive negative thoughts, and (2) improvement of the affective valence associated to self-referential adjectives, and that these changes will be associated with decreased connectivity between structures mentioned above. The present early feasibility study is an initial step that aims to determine its feasibility and help with the planning of a larger study addressed at actual hypothesis testing.

DETAILED DESCRIPTION:
Depression represents a remarkable public health burden, accounting for a large amount of disability and societal costs, comparable to prevalent diseases in other areas of medicine. This is partly due to unsatisfactory outcomes of well-established therapies, including psychotropic drugs and different types of psychotherapy. As a response to this problem, therapeutics in psychiatry is moving from drug manipulation of neurotransmitter systems to modulation of brain circuits selectively involved in specific symptoms of depression. These efforts have been partially hampered, however, by heterogeneity of clinical manifestations in these disorders, such that different symptoms are hypothesized to be maintained by specific circuit-level dysfunctions, as well as by significant interindividual variation in those brain circuits, which calls for personalized approaches to achieve their successful modulation. Thus far, the efforts to accomplish individualized and precise modulation of aberrant circuits responsible for the expression of depression and anxiety symptoms have encountered three important, mutually related problems. First, widely available noninvasive neuromodulation techniques such as repetitive transcranial magnetic stimulation (rTMS) have poor spatial resolution and only reach superficial areas of the brain, which impedes the precise modulation of circuits that involve deep, minute subcortical gray matter structures and/or white matter connecting tracts. Second, surgical deep-brain stimulation procedures are more accurate but are too costly and risky to be implemented in any moderately sized proof-of-concept study at present. Third, it is unlikely that modification of the activity of a discrete brain circuit will target the entire complex behavioral macro of major depression. The investigators therefore chose to target a single measurable and replicable construct of depression, repetitive negative thinking (RNT). RNT is a transdiagnostic clinical manifestation that cuts across a variety of internalizing psychiatric disorders, but in the case of depression, it is associated with persistent symptoms, treatment resistance, proneness to relapse after treatment, and more suicidal ideation, behavior, and completed suicides. With the help of an emerging technology device recently acquired by LIBR, which can produce focused, reversible and noninvasive neuromodulation in deep brain structures (low-intensity transcranial focused ultrasound, tfUS), the investigators will probe the causal role of individually-identified circuits in the modulation of (a) the generation and maintenance of repetitive negative thinking (RNT), and (b) affective processing of self-referential adjectives. Specifically, the investigators will put to test the hypotheses that RNT and the affective load of self-referential adjectives can be improved by modulating components of an anteromedial brain circuit, identified on an individual basis as associated with high levels of RNT. Therefore, this project has two distinct phases. First, the investigators will use advanced structural-functional connectivity analysis techniques to define anatomical tracts that support functional connectivity alterations associated with high RNT. The investigators will refine and adjust results of whole-brain analyses, by focusing also on overlapping anatomical components of tracts pertaining to three well-established, historical psychosurgical targets of antidepressant and obsessional thinking treatment. Second, the investigators will employ the resulting regions of interest to inform the choice of the target(s) for tfUS neuromodulation, probing its effects on 1) neural processing of self-referential affective adjectives, 2) functional connectivity between regions known to have an anatomical connection in the individual participant, and 3) measures of RNT and clinical depression, including the degree of distress associated to the thought/s subjected to RNT. The investigators are in an ideal position to accomplish these objectives, given their experience with clinical management of these disorders, with the use of neuromodulation techniques, and expertise in the use of state-of-the-art structural and functional neuroimaging techniques, psychophysiological tools, and computational psychiatry methods.

ELIGIBILITY:
Inclusion Criteria:

1. Prior participation in the CoBRE study (WIRB Protocol #20182352) and selected as a component of the propensity-matched sample of patients with major depression and varying intensities of RNT (in the form of Ruminative Response Scale (RRS) score; n=20), or healthy individuals with no psychiatric diagnosis (n=10), OR In the unexpected event that not enough participants can be recruited who meet criterion 1 (only 1 out of 6 studied patients would be incorporated into this study), participants will be newly recruited from newly recruited patients from the community or from the Mood and Anxiety Disorders inpatient unit at Laureate Psychiatric Hospital and Clinic.
2. A Patient Health Questionnaire (PHQ-9) score ≥ 10 at enrollment.
3. Provision of signed and dated informed consent form.
4. Subject provides verifiable contact information (name, telephone number(s), email and mailing address) for at least 2 persons who agree to be contacted by study personnel as deemed necessary.
5. Subject is followed by a licensed physician or a licensed mental health care provider (i.e., psychologist, LCSW) throughout study participation outside of LIBR.
6. Stated willingness to comply with all study procedures and availability for the duration of the study.
7. Male or female, aged 18 to 65 years.
8. In good current general health as evidenced by medical history.
9. Ability to comply with the study chronogram.
10. For females of reproductive potential: negative urine pregnancy screening test.

Exclusion Criteria:

1. Current use (within the last 30 days) of drugs of abuse or moderate / severe alcohol use disorder.
2. Lifetime diagnosis of schizophrenia spectrum disorder, other nonaffective psychotic disorders, or bipolar disorders.
3. Presence of cardiac pacemaker or any other MRI contraindication.
4. Pregnancy or lactation.
5. Febrile illness within the last two weeks.
6. Treatment with an investigational drug or participation in any other interventional research protocol in the last 2 weeks.
7. The participant is unable to understand the goal of the study, instructions, or the risks associated with the study as judged by a clinically trained assessment team member.
8. Clinical and/or imaging evidence of vascular, traumatic, or neurodegenerative disorders of the central nervous system (CNS), or other neurological disorders potentially compromising patient's participation in the study, or study results. This includes, but it is not limited to, any minor or major neurocognitive disorder including those caused by traumatic brain injury, Parkinson's disease, significant small-vessel disease, multiple sclerosis, Huntington's disease, early-onset Alzheimer's disease, chronic infections of the CNS or the meninges, previous chronic use of alcohol or CVA sequelae, or a Montreal Cognitive Assessment (MoCA) score <25 due to any cause. The PI can decide if a potential participant needs to be excluded due to some other cause of structural or functional compromise of the CNS (e.g., epilepsy).
9. Active suicidal ideation (as measured by Suicide-Risk-Assessment-C-SSRS "Yes" answers to items 3, 4 or 5 of Suicidal Ideation-Past 1 month section, or any "Yes" answer to any of the items of Suicidal Behavior-Past 3 months section), or any suicide attempt in the last year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Post-Sonication Change in the Intensity of Repetitive Negative Thinking | Pre- vs 10-minute post-sonication or sham intervention.
  Change of BSRI (Brief State Rumination Inventory) score; minimum value: 0, maximum value: 800; higher scores mean worse outcome.

SECONDARY OUTCOMES:
Suicide Safety Indicators | Pre- vs 1-hour and 1-week post-sonication or sham intervention.
  Change in Columbia-Suicide Severity Rating Scale (C-SSRS) score, minimum value: 0; maximum value: 25; higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsuchiyagaito A, Kuplicki R, Misaki M, Edwards L, Camprodon JA, Fitzgerald K, Khalsa SS, Philip NS, Paulus MP, Guinjoan SM. Reversible modulation of a deep white matter surgical target for depression with low-intensity focused ultrasound. Neuropsychopharmacology. 2026 Feb;51(3):612-621. doi: 10.1038/s41386-025-02252-7. Epub 2025 Sep 25. PMID 40999237